CLINICAL TRIAL: NCT05182372
Title: Enhancing Digital CBT-I to Improve Adherence and Reduce Disparities
Acronym: COACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Michigan (Other); National Jewish Health (Other)
Responsible Party: Principal Investigator, Philip Cheng, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14816
Record Dates: First submitted 2021-12-02; First posted 2022-01-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Insomnia
Keywords: digital CBTI; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Random assignment into experimental and control conditions at a 1:1 ratio
Who Masked: Investigator
Masking Description: The principle investigator will be blind to the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced dCBT-I (Experimental): This group will complete d-CBTI and be assigned a coach that will help with completion of the treatment and will be available to call personally to discuss questions and issues.
  Interventions: Behavioral: Enhanced dCBT-I
- Control dCBT-I (No Intervention): Participants in this group will complete dCBT-I individually without assistance from a healthcare provider

INTERVENTIONS:
Behavioral: Enhanced dCBT-I — Telehealth Coaching
  Arms: Enhanced dCBT-I

SUMMARY:
The primary objective of this research study is to increase adherence of Digital Cognitive Behavioral Treatment for Insomnia (dCBT-I). Additionally, this study will examine behavioral, physical, and sociocultural factors associated with treatment engagement.

DETAILED DESCRIPTION:
Insomnia is a debilitating condition that impacts one third of adults, with a majority not having access to proper treatment. Digital Cognitive Behavioral Treatment for Insomnia (dCBT-I). is a method that is becoming more accessible and with strong success rate with treatment completion; however, non-completion rates are common, specifically in those with low socioeconomic status (SES).

This study will examine the addition of telehealth coaching to dCBT-I to increase adherence rates. Telehealth coaching will aim to provide support to mitigate the impact of lower health literacy, and will also enhance self-efficacy as a mechanism to promote treatment persistence.

Participants will be recruited from the Henry Ford Health System (HFHS) outpatient network as well as the Medicare/Medicaid data warehouse. Subjects will be screened to determine eligibility, and then will be randomized into one of two insomnia treatment groups (control dCBT-I and dCBT-I with telehealth coaching). Treatment involves 6 weekly dCBT-I sessions. In the dCBT-I with coaching component, those who are at risk for treatment non-completion will be offered two telehealth sessions of brief behavioral therapy for insomnia. Those in the control dCBT-I who are at risk for treatment non-completion will be provided digital sleep education.

At the end of the treatment period, some participants will complete a semi-structured interview to assess for facilitators and barriers to treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* Determination of insomnia (ISI >14)

Exclusion Criteria:

* Age < 18
* Unwillingness/inability to participate
* Bipolar or Seizure Disorders
* Untreated sleep disorders other than insomnia
* Untreated and severe medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Risk of treatment non-completion | throughout the study until the final study visit, up to 6 weeks
  Determined based on missing two consecutive sessions of dCBT-I.Missing two consecutive sessions equals being behind on sessions by 14 days.
Treatment Completion | throughout the study until the final study visit, up to 6 weeks
  Completion of all 6 sessions of dCBT-I.
Adherence to Sleep Restriction | throughout the study until the final study visit, up to 6 weeks
  Determined based on the variance of sleep diary variables

SECONDARY OUTCOMES:
Insomnia | throughout the study until the final study visit, up to 6 weeks
  Insomnia Severity Index Score (0 to 28; higher scores correspond to worse severity)
Physical Environment | within 2 weeks of post-treatment
  Participants will be asked about the layout of their sleep environment as well as neighborhood characteristics. Sleep environment will be assessed using qualitative information on individual's surroundings and information such as their ability to adjust light levels, temperature, and sound. If it is easier for the individual to adjust these, then they have a better physical environment for sleep. Neighborhood characteristics will be evaluated with the Neighborhood Safety scale (scores range from 1 to 5; lower scores indicate more neighborhood safety).
Sociocultural environment | within 2 weeks of post-treatment
  Sociocultural environment is measured using a household roster and the Everyday Discrimination Scale. A household roster will ask participants to report the number of individuals in the household and characterize the relationship with the participant. No summary score exists for the household roster. The Everyday Discrimination Scale measures frequency of discrimination (scores range from 10 to 60; higher scores represent more frequent experiences of discrimination).

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Cheng, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Columbus Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No